CLINICAL TRIAL: NCT05447858
Title: Systematic Work Environment Model Incorporating Web-based Neck-specific Exercise for Dental Staff With Neck Pain: A Prospective Randomized Controlled Study (WorkCIT)
Brief Title: Systematic Work Environment Model Incorporating Web-based Neck-specific Exercise for Dental Staff With Neck Pain
Acronym: WorkCIT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of fundings
Sponsor: Linkoeping University (Other Government)
Collaborators: Ostergotland County Council, Sweden (Other); Lund University (Other); Karlstad University (Other); The University of Queensland (Other); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Anneli Peolsson, Professor, PhD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2022-02188-02
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Workplace; Neck Pain; Exercise
Keywords: Neck pain; Workplace; Counseling; Exercise; Internet; Cervical spine
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomization will be handled by a person not involved in intervention or evaluation. Investigators/ assessors will be blinded for randomization.
  This is a prospective, longitudinal, randomised, controlled multi-centre trial with two parallel treatment arms and blinded investigators conducted according to a detailed protocol. A total of 240 employees with WRNP will be recruited. The main outcome is neck pain intensity. Secondary outcomes are work ability, function, health-related quality of life, work absenteeism, work-related factors, work adjustments made. Cost-effectiveness will be studied if significant differences appear between randomization groups regarding health-related quality of life and will in that case be reported in a separate paper.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managerial support in using systematic work environment evaluation and adjustment (SWEA) (Active Comparator): Managerial support in using SWEA and the Prehab guide to enhance employees' work situation. Individual work adaptations are adaptations to everyone´s ability in the physical, organisational, and social work environment that aim to enable an employee with reduced ability to perform the normal work, continue working, or plan for a sustainable return to work. The Prehab guide contains a self-assessment test for the employee based on the requirements of the work and one's own ability that can be used in the dialogue with the manager. It also contains suggestions for activities to create a healthier workplace, such as discovering early signals of stress or pain, creating a caring workplace culture and boundaries, regular contact with an employee that is on sick-leave, clear and established safety procedures and routines for the work environmental work, routines for cooperation with other parties, and to learn from one's own and colleague's experiences in an open, permissive climate.
  Interventions: Other: Neck-specific exercise
- Neck-specific exercise in addition to SWEA (Experimental): NSEs will be performed based on a well-structured framework of evidence-based exercises for facilitation of deep neck muscles, improved interaction between the different muscle layers of the neck, increased neck muscle endurance, and improved postural control [15, 30]. To ensure that the exercises are learned and performed correctly, the participant will meet with a physiotherapist a total of four times, once during weeks 2, 3, 4, and 7 (week 1=first visit for a clinical examination due to law) for instruction, guidance, and support. In addition to photos, videos, and text regarding the exercises, the digital support (web-based program at the support and treatment platform Inera via 1177 managed by the County Councils) also contains information about why it is important to exercise the neck muscles, factors that may cause neck pain, how relapses can be handled, ergonomic advice related to the neck, and an exercise diary.
  Interventions: Other: SWEA

INTERVENTIONS:
Other: SWEA — Managers with one or several l staff experiencing WRNP will be educated in the Prehab guide. The manager should read and listen to all modules and a 1-h lecture recorded by the research team before participating in two workshops (4 h each), together with other managers and an experienced expert in work environmental health and rehabilitation. In the workshops, different themes will be discussed, such as physical, psychological, and organisational work-related health, prevention, and rehabilitation, how to lead problem-solving dialogue, how work-related adaptations can be performed related to WRNP, and questions about the Prehab guide. The Prehab guide will be used to deliver managerial support in the work with the Swedish Work Environment Authority's regulations regarding SWEA and the prevention of ill health, sick leave, and accidents, work adaptations, and workplace-oriented rehabilitation.
  Arms: Neck-specific exercise in addition to SWEA
Other: Neck-specific exercise — NSEs will be performed based on a well-structured framework of evidence-based exercises for facilitation of deep neck muscles, improved interaction between the different muscle layers of the neck, increased neck muscle endurance, and improved postural control .
  Arms: Managerial support in using systematic work environment evaluation and adjustment (SWEA)

SUMMARY:
The aim of study; WorkCIT is to investigate whether managerial support in using systematic work environment evaluation and adjustment (SWEA) with/without additional 3 month web-based NSEs with four visits to a physiotherapist is effective in promoting reduced neck pain and disability among dental health care professionals (DHCP) with work-related neck pain (WRNP).

The aim of the subgroup studies is to investigate biomarkers and tissue changes and the association with pain, work ability, and other outcomes before and after SWEA with or without NSEs. Furthermore, to investigate dental staff experiences with the interventions and their impact on work ability, health and their work situation, and investigate managers experience of SWEA with support from the Prehab guide and workshops.

The hypothesis is that a combined effort with SWEA to promote the work situation together with NSEs will reduce neck pain intensity and improve work ability to a greater extent than the SWEA only.

Methods and analysis: This is a prospective, longitudinal, randomised, controlled multi-centre trial with two parallel treatment arms and blinded investigators conducted according to a detailed protocol following the guidelines in the CONSORT checklist. A total of 240 DHCP with WRNP will be recruited. The main outcome is neck pain intensity. Secondary outcomes are work ability, function, health-related quality of life, work absenteeism, work-related factors, and work adjustments made. Cost-effectiveness will be studied from a societal perspective if significant differences appear between randomization groups regarding health-related quality of life and will in that case be reported in a separate paper. To improve diagnostics and help assess the effectiveness of intervention biochemical sub-group studies will be performed before and after intervention to investigate pain related biomarkers. Interviews with a sub-group of participants and managers will be performed regarding work-ability, work adjustments and experiences of interventions.

DETAILED DESCRIPTION:
Introduction: Neck pain among dental health care professionals (DHCP) is a growing societal problem. It is compulsory by law, for managers to work with systematic work environment evaluation and adjustment (SWEA), though managers knowledge of this approach is often deficient. Managerial support in using SWEA to enhance employees' work situation has not been investigated in regards to work-related neck pain (WRNP). Clear guidelines on interventions for WRNP are lacking. Neck-specific exercise (NSE) is the method with the most evidence regarding treatment for neck problems in general but has not been investigated for WRNP. The aim of study; WORKCIT is to investigate whether managerial support in using SWEA with/without additional 3 month web-based NSEs with four visits to a physiotherapist is effective in promoting reduced neck pain and disability among DHCP with WRNP. More specifically, the main project aims to: Compare the effects of SWEA with a focus on adjustments at work and support for DHCP (aimed for all staff) by their manager with the addition (half of the staff) of an E-health solution of NSEs in combination with four visits to a physiotherapist with regards to neck pain intensity, disability, work ability, health, and cost-effectiveness; Investigate whether a participatory approach of workshops and digital education for managers in SWEA/ Prehabguiden Suntarbetsliv (Prehab guide) enhance the work environment (organisational, social, and physical), including individual support and adjustment of the work situation, reducing their neck pain intensity; Investigate if NSE reduces WRNP in addition to SWEA; Identify underlying factors associated with the outcome following work interventions with or without exercise regarding pain, work ability, and health.

The aim of the subgroup studies is to investigate biomarkers and tissue changes and the association with pain, work ability, and other outcomes before and after SWEA with or without NSEs. Furthermore, to investigate dental staff experiences with the interventions and their impact on work ability, health and their work situation, and investigate managers experience of SWEA with support from the Prehab guide and workshops.

The hypothesis is that a combined effort with SWEA to promote the work situation together with NSEs will reduce neck pain intensity and improve work ability to a greater extent than the SWEA only.

Methods and analysis: This is a prospective, longitudinal, randomised, controlled multi-centre trial with two parallel treatment arms and blinded investigators conducted according to a detailed protocol following the guidelines in the CONSORT checklist. A total of 240 DHCP with WRNP will be recruited. The main outcome is neck pain intensity. Secondary outcomes are work ability, function, health-related quality of life, work absenteeism, work-related factors, and work adjustments made. Cost-effectiveness will be studied from a societal perspective if significant differences appear between randomization groups regarding health-related quality of life and will in that case be reported in a separate paper. To improve diagnostics and help assess the effectiveness of intervention biochemical sub-group studies will be performed before and after intervention to investigate pain related biomarkers. Interviews with a sub-group of participants and managers will be performed regarding work-ability, work adjustments and experiences of interventions.

Ethics and dissemination: The study is approved by the Swedish Ethical Review Authority. The processing of personal data according to the General Data Protection Regulation will be registered at Linköping University before the start of the study. The results will be published in scientific journals, presented at scientific conferences and in meetings with caregivers, disseminated in lectures to the medical faculty and patient associations, and communicated in the media.

ELIGIBILITY:
Inclusion Criteria:

For employees:

* Self-reported WRNP lasting at least 4 weeks
* Current neck pain ≥ 3 on the numeric rating scale (Numeric Rating Scale (NRS), 0-10)
* Working age, 18-65 y
* Neck problems clinically verified by clinical examination to ensure study criteria are met
* Answered the baseline questionnaire and attended the first intervention visit
* Completed and signed informed consent, including approval, to contact their immediate supervisor regarding work adaptations.

For managers:

• Being a head/ manager of a dental clinic.

Exclusion Criteria:

Red flags and illness/injury that are contraindicated for or hinder exercise or may be confounding factors for the results including:

* Known pregnancy
* Cannot understand/communicate in Swedish and would be unable to understand information about the study or answer questionnaires.

For blood samples (not wanting to participate does not constitute exclusion from the RCT), the following exclusion criteria are added:

• Increased tendency to bleed and use of blood thinners.

For the microdialysis subgroup (n=30), consecutively asked, 15 persons/group; not wanting to participate does not constitute exclusion from the RCT), the following exclusion criteria are added:

* Cannot imagine refraining from anti-inflammatory drugs (NSAIDs) during the 2 days prior to microdialysis
* Hypersensitivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Current neck pain intensity | Change in current neck pain intensity from baseline, to 3 month (after intervention) and until the 15 month follow-up (1 year after intervention ended).
  Current neck pain intensity at 15 months follow-up measured on the numeric rating scale (NRS) (0=no pain and 10=worst imaginable pain)

SECONDARY OUTCOMES:
Work Ability Index (WAI) including Work Ability Scale (question no 1 in WAI) | Change in work ability from baseline to 3 month and 15 month follow-up
  Current work ability compared to when it was at its best, total score, between 7 and 49, poor (7-27), moderate (28-36), good (37-43) and excellent (44-49) work ability
Intensity of pain and bothersomeness | Change from baseline to 3 month and 15 month follow-up
  neck pain bothersomeness, headache intensity on NRS
Frequency of pain, symptoms and medications | Change from baseline to 3 month and 15 month follow-up
  Frequency of pain, pain medication, neck stiffness, numbness/tingling into the arms, having problems lifting the arms, dizziness, sleep, concentration.
Neck specific function | Change from baseline to 3 month and 15 month follow-up
  Neck Disability Index, 0 to 50 points or 0 to 100%; 0= no disability
Symptom satisfaction | Change from baseline to 3 month and 15 month follow-up
  Symptom satisfaction; how patients would feel about having their current (the last 24-hours) neck symptoms for the rest of thir lives, 1=delighted, 7=terrible (according to Cherkin and Deyo)
Exercise/ Physical activity level | Change from baseline to 3 month and 15 month follow-up
  Exercise/ physical activity level, how much time do you spend a regular week doing physical exercise and regular physical exercise, respectively, in median minutes, more minutes= better
Health related quality of life, EQ-5D-5L | Change from baseline to 3 month and 15 month follow-up
  Euroqol 5 dimension; EQ-5D-5L, The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems, a summed score of all 5 questions will be used where 1=perfect health.
Perceived exertion at work | Change from baseline to 3 month and 15 month follow-up
  Borg scale of exertion, ratings of perceived exertion at work measured with the Borg scale; 0=no exertion, 10=major exertion
Sick-leave | Change from baseline to 3 month and 15 month follow-up
  sick leave numbers of days/month
Effort-Reward Imbalance | Change from baseline to 3 month and 15 month follow-up
  Effort-Reward Imbalance questionnaire, less than 1 is indicating a favour of rewards, more than 1 indicating a favour of effort
Risk identification at work | Change from baseline to 3 month and 15 month follow-up
  Structured multidisciplinary work evaluation tool, (SMET) will be used. The questionnaire asks about physically, environmentally and psychosocially demanding work items (30 items). A scale of 1-10 is used in the questionnaire, 1 is labeled "Not at all" and 10 is labeled "Highly".
Work adaptation | Change from baseline to 3 month and 15 month follow-up
  Open questions about work adaptation, such as self strategies to be able to work
Time sitting | Change from baseline to 3 month and 15 month follow-up
  Time sitting at work and during leisure time
Anxiety and depression | Change from baseline to 3 month and 15 month follow-up
  Hospital Anxiety and Depression Scale, 0-6= healthy, 7-10= mild to moderate, >10= (risk for/ indication of- a diagnos needs a clinical examination) anxiety or depression
Fullfilment of treatment expectation | Change from baseline to 3 month and 15 month follow-up
  Fullfilment of treatment expectation, have your expectations been fullfilled, yes, yes partly, no
Overall outcome | Cross-sectional 3 month and 15 month follow-up
  Global rating of change scale, -5= much worse, 0= unchanged, 5=much better/restored
Satisfaction with the caregiver visits in the study | Cross-sectional 3 month and 15 month follow-up
  Patient enablement questionnaire, The PEI is a 6-item scale that has been used in general prac-tice to evaluate quality of care. The highest possible score is 12, with higher scores indicating greater enablement.
Cost-effectiveness. (Will be analysed in a later stage if differences appear between groups) | From the time period between baseline to 15 month follow-up
  Through calculation of direct costs; quantity and type of care (inside and outside the study also including drugs related to pain) from registers and from questionnaires, indirect costs; mainly production loss from registers and from questionnaire. Will be calculated if there is a difference between randomisation groups and will in that case be presented in a paper of its own.
Saliva samples and blood samples (Sub-group, not in the RCT) | Change from baseline to 3-month follow-up in the subgroup of the RCT population
  Experimental sub-group study. Protein analysis to investigate differences between patients and healthy controls, biomarkers of inflammation and stress. Will be performed in a sub-group. Saliva will be collected with Salivette. Venous blood samples (10-20 ml) from the elbow fold will be collected in EDTA tubes. Identification and quantification of proteins. In a subgroup of the RCT population. Comparisons will be made with healthy controls. Permits for biobank is available.
Microdialysis, tissue changes in the middle of Trapezius (Subgroup study, not in the RCT) | Change from baseline to 3 month, subgroup of the RCT population
  Biomechanical changes interstitialli in M. Trapezius. Through microdialysis technology, it is possible to monitor biochemical changes interstitially in the tissue. The technique involves the exchange of substances via diffusion between the tissue and a diaphragmatic cateter inserted into the tissue and flushed by a fluid (perfusate) that is similar in chemical composition to the fluid in the muscle interstitium. Comparisons will be made with healthy controls.
Interview study of employees (Sub-group study, not in the RCT) | after intervention fulfilled, sub-group of the RCT population, n=approximately 15
  Employees experience with interventions and their impact on work ability, health and work situation. Sub-group of the RCT population.
Interview with managers (Subgroup study) | After having at least one employee participating and fulfilled the study.
  Interview with managers regarding the experience of using SWEA and the Prehabguide. A subgroup will be interviewd, Approximately n=approximately 15.
Perceived work environment problems | Description and change from baseline to 3 month and 15 month follow-up
  During the past 7 days, how much did your work environment-related problemsaffect your performance at work? A scale 0 - 10 is used, 0 is labeled " Workenvironment problems have not affected my work performance" and 10 is labeled"Work environment problems completely prevented me from working". A higher score indicates a worse outcome.
Work environment related production loss | Description and change from baseline to 3 month and 15 month follow-up
  During the past 7 days, how much did your work environment-related problemsaffect your performance at work? A scale 0 - 10 is used, 0 is labeled " Workenvironment problems have not affected my work performance" and 10 is labeled"Work environment problems completely prevented me from working". A higherscore indicates a worse outcome.
Self-rated work situation regarding neck position at work | Description and change from baseline to 3 month and 15 month follow-up
  Numeric rating scale 0-10, 10= very satisfied
Health related quality of life, EQ thermometer | Change from baseline to 3 and 15 months
  Euroqol vertical visual analogue scale, 0-100, 100=perfect health

OTHER OUTCOMES:
Profession | Baseline
  Swedish standard for work classification
Background data | Baseline
  Age, sex, education, family situation, pain duration, expectations, smoking history
Treatment outside the study | Descripton baseline, 3 month, 15 month
  A in-house made question about treatment outside the study at different health care professionals, number of visits and if better or unchanged and earlier treatment for neck pain before inclusion into the study
Profession | Description baseline, 3 month and 15 month
  Open question of profession
work situation | Descriptive data at baseline, 3 month and 15 month follow-up
  Description of occupation, work tasks, type of employer, working hours, years in occupation, in-house made questions as basic background information to understand each workers work situation and change in work sitiation

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, Prof., PhD, Principal Investigator — Linkoeping University

IPD SHARING:
Plan to Share IPD: No
The data is protected by the Swedish health secrets act and the European General Data Protection Regulation. Data will be presented on a group level without possibility for individual identification.